CLINICAL TRIAL: NCT01286675
Title: A Pilot Study to Evaluate the Effect of Eltrombopag Plus G-CSF on Human CD34+ Cell Mobilization and Ex Vivo Colony Proliferative Capacity in Patients With Multiple Myeloma Undergoing Autologous Stem Cell Transplantation
Brief Title: Effect of Eltrombopag Plus G-CSF on Human CD34+ Cell Mobilization in Multiple Myeloma Patients Undergoing ASCT
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Dana-Farber Cancer Institute (Other)
Responsible Party: Principal Investigator, Nancy Berliner, MD, Chief, Division of Hematology, Dana-Farber Cancer Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 10-346
Record Dates: First submitted 2011-01-28; First posted 2011-01-31 (Estimated); Last update posted 2019-03-01 (Actual); Status verified 2019-02

CONDITIONS: Multiple Myeloma
Keywords: ASCT; G-CSF
MeSH Terms: conditions — Multiple Myeloma | interventions — eltrombopag

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Eltrombopag (Experimental): 0 mg Eltrombopag
  Interventions: Drug: Eltrombopag

INTERVENTIONS:
Drug: Eltrombopag — oral eltrombopag, 50 mg, 100 mg, 150 mg, days 2-15
  Other Names: SB-497-115-GR

SUMMARY:
Eltrombopag may improve the cell collection available for Autologous Stem Cell Transplant(ASCT). The overall goal is to determine if adding Eltrombopag to the standard ASCT will increase the number of blood cells collected and reduce the number of times blood needs to be collected. This study will also determine the highest dose of Eltrombopag that can be used without causing serious side effects.

DETAILED DESCRIPTION:
Subjects will receive standard treatment for autologous stem cell transplant. Subjects will be assigned to receive no Eltrombopag or one of three dose levels of Eltrombopag. Subjects will receive oral Eltrombopag on days 2-15 of treatment.

ELIGIBILITY:
Inclusion Criteria:

* Multiple myeloma
* Stable or responsive disease after at least 2 cycles of conventional chemotherapy
* Slated to undergo autologous peripheral blood stem cell transplant
* Normal organ and marrow function

Exclusion Criteria:

* Myocardial infarction within 6 months of treatment
* Receiving other study agents
* Pregnant or breastfeeding
* Uncontrolled intercurrent illness
* Evidence of active or recent history of thromboembolic disease
* Previous history of primary platelet disorder or bleeding disorder
* History of a different malignancy unless disease free for at least 5 years

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2011-03; Primary Completion 2016-12 (Actual); Study Completion 2018-12 (Actual)

PRIMARY OUTCOMES:
Evaluate the median fold increase in the number of CD34+ cells/kg mobilized at each dose level. | 1 year
  Evaluate the median fold increase in the number of CD34+ cells/kg mobilized at each dose level.
Evaluate the number of apheresis procedures required to obtain at least 2 x 10^6 CD34+ cells/kg at each dose level | 1 year
  Evaluate the number of apheresis procedures required to obtain at least 2 x 10^6 CD34+ cells/kg at each dose level
Determine the maximum tolerated dose of eltrombopag with granulocyte colony-stimulating factor. | 1 year
  Determine the maximum tolerated dose of eltrombopag with granulocyte colony-stimulating factor.

SECONDARY OUTCOMES:
Evaluate the median fold increase in platelet counts at each of the dose levels | 1 year
  Evaluate the median fold increase in platelet counts at each of the dose levels
Evaluate the median fold increase in hematopoietic colony forming capacity of CD34+ cells at each dose level | 1 year
  Evaluate the median fold increase in hematopoietic colony forming capacity of CD34+ cells at each dose level

CONTACTS AND LOCATIONS:
Overall Officials: Nancy Berliner, MD, Principal Investigator — Dana-Farber Cancer Institute
Locations (1):
- Dana Farber Cancer Institute, Boston, Massachusetts, United States